CLINICAL TRIAL: NCT04019275
Title: ENGAGE Pilot Study: Promoting Participation and Health After Stroke
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The COVID pandemic impeded recruitment at two sites (Pitt 80% target recruitment, Wash U 70% target recruitment) and prohibited recruitment at one site (UIC). Study was terminated when funding was spent.
Sponsor: University of Pittsburgh (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Elizabeth R. Skidmore, PhD, OTR/L, Professor, Occupational Therapy, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO19030256; UL1TR001857 (NIH); UL1TR002345 (NIH)
Record Dates: First submitted 2019-07-11; First posted 2019-07-15 (Actual); Results first posted 2023-06-23 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: disability, rehabilitation
MeSH Terms: conditions — Stroke | interventions — engage 8200

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ENGAGE (Experimental): The intervention blends social learning, guided discovery, and skill training to promote community participation after stroke. The intervention is delivered in a group format and comprises group learning activities and individual action planning activities that address barriers to community participation after stroke.
  Interventions: Behavioral: ENGAGE

INTERVENTIONS:
Behavioral: ENGAGE — ENGAGE blends social learning, guided discovery and skill training focused on community participation

SUMMARY:
This is a multi-site single-arm community-based pilot study examining the feasibility, acceptability, safety, and estimated effects of the ENGAGE intervention, a community-based intervention to promote community participation after stroke. The study will also characterize variances in changes in community participation outcomes. These findings will provide the pilot data needed to inform a multi-site randomized controlled clinical trial.

DETAILED DESCRIPTION:
Significant advancements in acute medical management have shifted stroke from an acute condition with a high prevalence of mortality to a chronic condition with high prevalence of morbidity. One of the leading causes of chronic illness and disability worldwide, stroke results in residual sensorimotor, cognition, and communication impairments. These impairments reduce over time, but few people have complete restoration of function. Hence, people with stroke-related disability do not resume pre-stroke levels of community participation (education; paid or volunteer work; civic, social, and religious activities; and leisure). Low levels of community participation are associated with inactivity, sedentary behavior, and social isolation, each contributors to cardiovascular disease, diabetes, obesity, pulmonary conditions, depression - and secondary stroke. These consequences are particularly problematic for people with low income who have limited resources.

Investigators at the University of Pittsburgh, Washington University, and the University of Illinois at Chicago have designed a self-management training program that uses social learning, motivational interviewing, and guided discovery to help people with mild to moderate stroke-related disability resume community participation, and to develop a strong network of social support. However, the combination of these elements has yet to be studied in people with chronic stroke-related disability who live with low income - one of the most vulnerable segments of the population. By partnering with the Community Research Fellows Program at Washington University and the Community PARTners Program at the University of Pittsburgh, this multi-site team seeks to design and implement a culturally-responsive program to promote community participation among people with stroke-related disability and low income. This new collaboration is the next logical step in the development and examination of community-based interventions to promote self-management and community participation after stroke.

The overall purpose of this research study is to examine the feasibility, safety, and acceptability of a multi-site community-based intervention to promote self-management of community participation after stroke, with a particular focus on the needs of people with low income. The study will also characterize variances in intervention response.

ELIGIBILITY:
Inclusion Criteria:

* ages 18 and older
* chronic stroke (minimum 3 months)
* community-dwelling
* mild to moderate stroke-related disability (NIHSS<=16)
* restrictions in community participation (ACS <80% of pre-stroke activities)
* low income (uninsured or underinsured)
* able to provide written informed consent

Exclusion Criteria:

* currently receiving rehabilitation serves
* dementia diagnosis
* severe aphasia (BDAE=0 or 1)
* current major depressive disorder (unless treated and in partial remission)
* current bipolar or psychotic disorder
* substance abuse within 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-12-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth R Skidmore, PhD, Principal Investigator — University of Pittsburgh; Carolyn Baum, PhD, Principal Investigator — Washington University School of Medicine; Joy Hammel, PhD, Principal Investigator — University of Illinois at Chicago
Locations (3):
- United States (3):
  - University of Illinois at Chicago, Chicago, Illinois
  - Washington University, St Louis, Missouri
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 38 participants provided informed consent and were eligible for the study. 8 participants withdrew before starting intervention (3 due to scheduling, 3 due to difficulty with accessing technology for the intervention, 1 was hospitalized, 1 withdrew at family request). 30 participants started the protocol.
Period: Overall Study
Arm/Group | ENGAGE
Started | 30
Completed | 24
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | ENGAGE
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.28 (12.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
PROMIS Ability to Participate in Social Roles [Mean (Standard Deviation); unit: T-score] — The PROMIS Ability to Participate in Social Roles scale measures difficulty participating in social roles and activities. Eight items are rated on a Liker-type scale from 1=always having difficulty to 5=never having difficulty. Raw total scores (range 8 to 40) are converted to standardized T-scores with a population mean of 50, with a standard deviation of 10. Higher T-scores are associated with less difficulty. A T-score of 40 is considered subclinical difficulty with ability to participate in social roles and activities.
  T-score | 43.48 (7.34)

OUTCOME MEASURES:

1. Primary Outcome: Fidelity, Indicated by Score of 18 or Higher Out of 20 on the ENGAGE Fidelity Checklist
Description: number of sessions attaining >= 90% adherence to protocol; an independent evaluator will assess a random 20% of sessions using the ENGAGE Fidelity Checklist; the Checklist has 20 items, each rated as 2=exceptional, 1=adherent, 0=not adherent
Time Frame: week 7
Population: Fidelity was observed for 4 randomly selected sessions from 24 total session, or 17% of group sessions involving 9 participants. After this point, fidelity assessment was halted due to the COVID pandemic.
Measure: Number; unit: sessions
Units Other Than Participants: sessions
Arm/Group | ENGAGE
Number analyzed (Participants) | 9
Number analyzed (sessions) | 4
sessions | 4

2. Primary Outcome: Acceptability, Indicated by Score 24 or Higher Out of 32 on the Client Satisfaction Questionnaire
Description: Number of participants attaining >= 90% satisfaction; satisfaction is rated on 8 items with a 4-point Likert-type scale, 4 indicating very high satisfaction. Items are summed with total score ranging from 8 indicating poor satisfaction to 32 indicating very high satisfaction.
Time Frame: week 7
Population: One participant did not complete the Client Satisfaction Questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | ENGAGE
Number analyzed (Participants) | 23
Participants | 20

3. Primary Outcome: Adverse Events, Defined as Reported Injuries or Injurious Falls
Time Frame: week 7
Measure: Count of Participants; unit: Participants
Arm/Group | ENGAGE
Number analyzed (Participants) | 24
Participants | 0

4. Secondary Outcome: Cohen's d Effect Size of the Change From Week 1 to Week 7 in PROMIS Ability to Participate in Social Roles
Description: The PROMIS Ability to Participate in Social Roles scale measures difficulty participating in social roles and activities. Eight items are rated on a Liker-type scale from 1=always having difficulty to 5=never having difficulty. Raw total scores (range 8 to 40) are converted to standardized T-scores with a population mean of 50, with a standard deviation of 10. Higher T-scores are associated with less difficulty. A T-score of 40 is considered subclinical difficulty with ability to participate in social roles and activities.
  A Cohen's d=.20 is considered a small effect size, d=.50 is considered a medium effect size, and d=.80 is considered a large effect size. A positive Cohen's d effect size indicates a higher score at week 7 than week 1. A negative Cohen's d effect size indicates a higher score at week 1 than week 7.
Time Frame: week 1 vs week 7
Measure: Number (95% Confidence Interval); unit: Cohen's d effect size
Arm/Group | ENGAGE
Number analyzed (Participants) | 24
Cohen's d effect size | 0.38 [-0.11 to 0.94]

ADVERSE EVENTS:
Time Frame: 7 weeks
Arm/Group | ENGAGE
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

LIMITATIONS AND CAVEATS:
The ENGAGE Fidelity Checklist was not finalized due to changes in procedures during the COVID pandemic. Thus, while 4 of 24 sessions involving 9 participants were assessed for fidelity, and all 4 sessions met criteria for fidelity, the method for assessing fidelity was still in development and was only applied to a limited sample of sessions. Data pertaining to this should be interpreted with caution.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-05-28): https://cdn.clinicaltrials.gov/large-docs/75/NCT04019275/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-16): https://cdn.clinicaltrials.gov/large-docs/75/NCT04019275/ICF_000.pdf